CLINICAL TRIAL: NCT00143416
Title: Long-Term Study of B2036-PEG in Acromegaly - Long Term Study With B2036-PEG -
Brief Title: Long Term Study With B2036-PEG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6291011
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — pegvisomant

INTERVENTIONS:
Drug: Pegvisomant

SUMMARY:
Primary objective: To investigate the efficacy and safety of Pegvisomant in Japanese patients with acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acromegaly who have received at least one dose of B2036-PEG in the preceding study (A6291009).

Exclusion Criteria:

* Switching to other therapeutic methods for acromegaly

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2004-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of long-term B2036-PEG therapy in patients with acromegaly

SECONDARY OUTCOMES:
PK/PD evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Japan (8):
  - Pfizer Investigational Site, Kobe, Hyogo PREF
  - Pfizer Investigational Site, Kozukue-cho, Kouhoku-ku, Yokohama-shi, Kanagawa
  - Pfizer Investigational Site, Kyoto, Kyoto
  - Pfizer Investigational Site, Hamamatsu, Shizuoka
  - Pfizer Investigational Site, Bonkyo-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo
  - Pfizer Investigational Site, Gakuhara, Kishiwada, Osaka
  - Pfizer Investigational Site, Sannomaru-cho, Naka-ku, Nagoya-shi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6291011&StudyName=Long%20Term%20Study%20with%20B2036-PEG